CLINICAL TRIAL: NCT01643070
Title: Randomized Phase II Trial of Preoperative Chemoradiation With or Without Induction Chemotherapy In Patients With Locally Advanced Or Borderlinely Resectable Rectal Cancer With Resectable Synchronous Liver Metastases
Brief Title: Preoperative CRT With or Without Induction Chemotherapy for Rectal Cancer With Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: XELOX-RT
Record Dates: First submitted 2011-11-01; First posted 2012-07-17 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer; Liver Metastases
Keywords: Rectal cancer; Liver metastases; Capecitabine; Oxaliplatin
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX RT (Active Comparator): Concurrent XELOX-RT (Capecitabine, Oxaliplatin, radiotherapy)
  Interventions: Drug: Capecitabine, Oxaliplatin; Radiation: Radiotherapy
- Induction XELOX (Active Comparator): Induction XELOX(Capecitabine, Oxaliplatin) followed by XELOX-RT (Capecitabine, Oxaliplatin, radiotherapy)
  Interventions: Drug: Capecitabine, Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin — Induction chemotherapy - Induction XELOX (Capecitabine 1250 mg/m2 PO twice daily on D1-14 and oxaliplatin 130 mg/m2 on D1, every 3 weeks for 2 cycles) Preoperative chemoradiotherapy - XELOX RT (Capecitabine 825 mg/m2 PO twice daily during radiotherapy and oxaliplatin 50 mg/m2/day on weekly.)
Radiation: Radiotherapy — Preoperative radiotherapy, 5040 cGy with 28 fractions

SUMMARY:
To investigate the feasibility of preoperative chemoradiation with oxaliplatin plus capecitabine, with or without prior induction chemotherapy in patients with locally advanced or marginally resectable rectal cancer with resectable synchronous liver metastases.

DETAILED DESCRIPTION:
Preoperative chemoradiation is now an initial treatment of choice for locally advanced resectable rectal cancer, and 5-fluorouracil is the standard agent during chemoradiation. Capecitabine is an oral fluoropyrimidine which has been thought to be a replacement for intravenous 5-fluorouracil, and several trials have proved that preoperative chemoradiation with capecitabine was also effective in this setting.

Oxaliplatin, a newer platinum agent, plus fluoropyrimidines (either 5-fluorouracil or capecitabine) is one of the standard cytotoxic chemotherapeutic regimen for metastatic colorectal cancer, and it is also proved to be effective as neoadjuvant chemotherapy for patients with liver only metastasis from colorectal cancer.

Approximately 25% of patients with colorectal cancer have liver metastases initially at the time of diagnosis and there have been quite well established evidences for clear survival benefits from hepatic metastasectomy in these patients. Treatment for colorectal liver metastases should be planned with consideration of both systemic chemotherapy and local treatment modality (surgery or radiofrequency ablation) because long term survival would be expected after curative liver metastasectomy. As mentioned previously, neoadjuvant oxaliplatin plus fluoropyrimidines before hepatic metastasectomy improved disease-free survival, thus it is thought to be that better systemic controls would be achieved with perioperative oxaliplatin based chemotherapy.

In patients with locally advanced rectal cancer, preoperative chemoradiation with fluoropyrimidines improves local control but not systemic control. Recent randomized trials of preoperative chemoradiation with oxaliplatin plus fluoropyrimidines failed to show better local control rates than those with fluoropyrimidines alone. But it is too early to determine the non-superiority of preoperative chemoradiation with oxaliplatin plus fluoropyrimidines in terms of systemic control; long-term duration of follow-up is needed to determine the efficacy in terms of disease-free or overall survival and it is evident that oxaliplatin based chemotherapy is effective for systemic control in patients who will be candidate for liver metastasectomy.

Thus, the investigators planned a randomized phase II trial of preoperative chemoradiation with oxaliplatin plus capecitabine, with or without prior induction chemotherapy in patients with locally advanced or borderlinely resectable rectal cancer with resectable synchronous liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum Tumor located within 12 cm from anal verge Clinical stage of T3-4 or N+ by rectal MRI ± endorectal ultrasound Age over 18 years No prior systemic treatment or radiation Adequate major organ functions Borderline resectability of primary rectal cancer Complete resectability of liver metastases (measurable by RECIST 1.1)

Exclusion Criteria:

* Unresectable liver metastases (6 or more metastatic lesions, major vessel invasion)
* Extrahepatic metastasis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2010 and May 2014, a total of 38 patients from 3 centers in Korea were enrolled. They underwent random assignment and 18 patients were assigned to arm A and 20 to arm B. The cutoff date for this report was March 15, 2015. Baseline characteristics of these patients are presented in Table 1, and they were well balanced between the 2 arms. The median number of LM was 2 and cT3N+ was the most common clinical disease stage in both arms.
Groups:
- Induction XELOX: Induction XELOX followed by XELOX-RT
  Capecitabine, Oxaliplatin: Induction chemotherapy - Capecitabine (1250 mg/m2 PO twice daily on D1-14 and oxaliplatin 130 mg/m2 on D1, every 3 weeks for 2 cycles) Preoperative chemoradiotherapy - Capecitabine 825 mg/m2 PO twice daily during radiotherapy and oxaliplatin 50 mg/m2/day on weekly.
  Radiotherapy: Preoperative radiotherapy, 5040 cGy with 28 fractions
- XELOX RT: Concurrent XELOX-RT
  Capecitabine, Oxaliplatin: Induction chemotherapy - Capecitabine (1250 mg/m2 PO twice daily on D1-14 and oxaliplatin 130 mg/m2 on D1, every 3 weeks for 2 cycles) Preoperative chemoradiotherapy - Capecitabine 825 mg/m2 PO twice daily during radiotherapy and oxaliplatin 50 mg/m2/day on weekly.
  Radiotherapy: Preoperative radiotherapy, 5040 cGy with 28 fractions
Period: Overall Study
Arm/Group | Induction XELOX | XELOX RT
Started | 18 | 20
XELOX-RT Received | 15 | 0
Underwent Surgery | 16 | 19
Completed (Received adjuvant XELOX) | 14 | 17
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 1 | 0
Not completed — Pregressive disease | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Induction XELOX-RT (Arm A): induction XELOX followed by XELOX-RT (arm A)
- XELOX-RT Alone (Arm B): no induction XELOX, XELOX-RT alone (arm B)
- Total: Total of all reporting groups
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B) | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Customized [Median (Full Range); unit: years]
  Age (years), median (range) | 60 [32 to 73] | 56 [37 to 76] | 58 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 15 | 19 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Perfomance status (ECOG PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale 0=Fully active, able to carry on all pre-disease performance without restriction;
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;
  Participants
    0 | 0 | 5 | 5
    1 | 18 | 15 | 33
Distance of the primary tumor from the anal verge [Count of Participants; unit: Participants]
  ≤ 4 cm | 6 | 13 | 19
  > 4 and ≤ 8 cm | 10 | 7 | 17
  > 8 cm | 2 | 0 | 2
Tumor differentiation [Count of Participants; unit: Participants]
  Well differentiated | 3 | 3 | 6
  Moderately differentiated | 13 | 16 | 29
  Poorly differentiated/signet ring cell/mucinous | 0 | 1 | 1
  Undetermined | 2 | 0 | 2
Clinical T Stage [Count of Participants; unit: Participants] — Clinical staging determines how much cancer there is based on rectal magnetic resonance imaging (MRI). The T element designates the size and invasiveness of the primary tumor.
  cT3=Tumor invades through the muscularis propria into pericolorectal tissues; cT4=Tumor penetrates to the surface of the visceral peritoneum or directly invades or adheres to other organs or structures
  Participants
    cT3 | 12 | 16 | 28
    cT4 | 6 | 4 | 10
Clinical N Stage [Count of Participants; unit: Participants] — Clinical staging determines how much cancer there is based on rectal magnetic resonance imaging (MRI). The N element designates the extent of regional lymph node involvement.
  cN0=No regional lymph node metastasis; cN1=One to Three regional lymph nodes are positive (tumor in lymph nodes measuring ≥0.2mm), or any number of tumor deposits are present and all identifiable lymph nodes are negative; cN2=Four or more regional nodes are positive;
  Participants
    cN0 | 1 | 0 | 1
    cN1 | 5 | 5 | 10
    cN2 | 12 | 15 | 27
Number of liver metastases [Count of Participants; unit: Participants]
  1 metastases | 6 | 7 | 13
  2 metastases | 4 | 5 | 9
  ≥3 metastases | 8 | 8 | 16
Number of liver metastases [Count of Participants; unit: Participants]
  1 | 6 | 7 | 13
  2 | 4 | 5 | 9
  ≥3 | 8 | 8 | 16
Largest size of liver metastases (cm), median (range) [Median (Full Range); unit: cm] | 1.8 [1.0 to 7.4] | 2.4 [1.0 to 6.9] | 2.1 [1.0 to 7.4]
Carcinoembryonic antigen (ug/ml), median (range) [Median (Full Range); unit: ng/ml] | 7.4 [0.7 to 548.0] | 6.9 [1.4 to 219.0] | 7.15 [0.7 to 548.0]

OUTCOME MEASURES:

1. Primary Outcome: Quality of Surgery for Primary Tumor
Description: R0 = complete resection with grossly and microscopically negative margins of resection; R1 =grossly negative but microscopically positive margins of resection; R2 = grossly and microscopically positive margins of resection
Time Frame: Arm A = Induction chemotherapy (XELOX, 6 weeks) followed by chemoradiotherapy (XELOX plus radiotherapy) to surgery (6 weeks); Arm B = Chemoradiotherapy (XELOX plus radiotherapy) to surgery (6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B)
Number analyzed (Participants) | 18 | 20
Participants
  Surgery not performed | 2 | 1
  R0 | 15 | 19
  R1 | 1 | 0
Statistical Analysis 1: Comparison: Induction XELOX-RT (Arm A) vs XELOX-RT Alone (Arm B); Test type: Superiority; p = 0.719, t-test, 1 sided; Odds Ratio (OR) = 1.500, 95% CI 2-sided [0.346 to 6.501]

2. Primary Outcome: Quality of Surgery for Liver Metastases
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B)
Number analyzed (Participants) | 18 | 20
Participants
  Surgery not performed | 2 | 1
  R0 | 11 | 12
  R0 with intraoperative Rdiofrequency ablation | 3 | 2
  R1 | 1 | 3
  R2 | 1 | 2

3. Primary Outcome: R0 Resection Rate of Both the Primary Tumor and Livermetastases
Description: synchronous complete R0 resection rate, R0 = complete resection with grossly and microscopically negative margins of resection
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B)
Number analyzed (Participants) | 18 | 20
percentage of patients | 77.8 [58.6 to 97.0] | 70.0 [49.9 to 90.1]

4. Secondary Outcome: Pathologic Complete Response Rate of Primary Tumor
Description: The pathologic stage (ypT or N) was recorded according to the International Union Against Cancer TNM system. Pathologic complete response (ypCR) was defined as the absence of viable tumor cells in the surgical specimens, of the primary tumor (ypT0).
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B)
Number analyzed (Participants) | 18 | 20
percentage of participants | 11.1 [0 to 25.6] | 5.0 [0 to 14.6]

5. Secondary Outcome: Tumor Regression Grade (Primary Tumor)
Description: The regression of the primary tumor was quantified according to the 5-point tumor regression grade proposed by Dworak.
  Complete regression = No tumor cells ; Near complete regression = Very few tumor cells; Moderate regression = Dominantly fibrotic changes with few tumor cells or groups; Minimal regression = Dominant tumor mass with obvious fibrosis
Time Frame: as for outcome 1
Population: Tumor regression grade (primary tumor)
Measure: Count of Participants; unit: Participants
Arm/Group | Induction XELOX-RT (Arm A) | XELOX-RT Alone (Arm B)
Number analyzed (Participants) | 18 | 20
Participants
  Surgery not performed | 2 | 1
  Total regression | 2 | 1
  Near total regression | 2 | 4
  Moderate regression | 10 | 11
  Minimal regression | 2 | 3

ADVERSE EVENTS:
Time Frame: Arm A = Induction chemotherapy (XELOX, 6 weeks) followed by chemoradiotherapy (XELOX plus radiotherapy) to surgery (6 weeks), followed by postoperative chemotherapy (XELOX, 18 weeks). Arm B = Chemoradiotherapy (XELOX plus radiotherapy) to surgery (6 weeks), followed by postoperative chemotherapy (XELOX, 18 weeks).
Description: Adverse events were analyzed by treatment exposure. This included Induction Chemotherapy (only Arm A), Preoperative Chemoradiotherapy, and Postoperative Chemotherapy
Groups:
- During Induction XELOX (Arm A): consisted of oxaliplatin 130 mg/m2 on day 1 and capecitabine 1000 mg/m2 twice daily on days 1 to 14, every 3 weeks for 2 cycles.
- During Preoperative Chemoradiotherapy With XELOX (Arm A); During Preoperative Chemoradiotherapy With XELOX (Arm B): consisted of radiation therapy with 45 Gy delivered in conventional fractionation (daily fractions of 1.8 Gy over a period of approximately 5 wk, excluding weekends) with or without additional 5.4 Gy delivery in daily fractions of 1.8 Gy over 3 days, oxaliplatin 50 mg/m2 weekly for 5 weeks, and capecitabine 825 mg/m2 twice daily on days 1 to 38 (during radiation therapy)
- During Postoperative XELOX (Arm A); During Posoperative XELOX (Arm B): Surgery was planned with total mesorectal excision and simultaneous liver metastasectomy with or without addition of radiofrequency ablation within 6 weeks after completion of preoperative treatments. Postoperative chemotherapy (postoperative CapeOx) consisted of oxaliplatin 130 mg/m2 on day 1 and capecitabine 1000 mg/m2 twice daily on days 1 to 14, every 3 weeks for 6 cycles.
Arm/Group | During Induction XELOX (Arm A) | During Preoperative Chemoradiotherapy With XELOX (Arm A) | During Preoperative Chemoradiotherapy With XELOX (Arm B) | During Postoperative XELOX (Arm A) | During Posoperative XELOX (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/15 | 0/20 | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/20 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 18/18 | 15/15 | 20/20 | 14/14 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | During Induction XELOX (Arm A) (N=18) | During Preoperative Chemoradiotherapy With XELOX (Arm A) (N=15) | During Preoperative Chemoradiotherapy With XELOX (Arm B) (N=20) | During Postoperative XELOX (Arm A) (N=14) | During Posoperative XELOX (Arm B) (N=17)
Leucopenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 7 | 9
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2 | 9 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 4 | 7 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 5 | 9 | 2 | 5
Nausea (Gastrointestinal disorders) | 6 | 3 | 7 | 4 | 9
Diarrhea (Gastrointestinal disorders) | 0 | 7 | 8 | 0 | 3
Sensory neuropathy (Nervous system disorders) | 9 | 5 | 13 | 14 | 14
Hand foot syndrome (Nervous system disorders) | 0 | 1 | 1 | 3 | 4
Anal pain (General disorders) | 1 | 4 | 8 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No